CLINICAL TRIAL: NCT04913246
Title: Comparison of the Triage Score With the Quick-Sofa Score (qSofa) in Septic Patients in the Emergency Department: Diagnostic and Prognostic Value.
Brief Title: Triage Score VS Quick-Sofa Score in Septic Patients in the Emergency Department
Acronym: Triage
Status: Completed | Type: Observational
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, PROFESSOR, Hôpital Universitaire Sahloul
Other Study IDs: Triage-Sepsis
Record Dates: First submitted 2021-05-25; First posted 2021-06-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Sepsis; Emergencies
Keywords: Sepsis; severity; prognosis; triage; Mortalty
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sepsis represents by its frequency, its morbidity and mortality and its cost to society a major public health issue with a constantly increasing incidence. It affects millions of people around the world each year and is the 2nd leading cause of death in intensive care units.

The incidence of sepsis has been estimated by the World Health Organization (WHO), based on US data, at 15 to 19 million cases of sepsis per year worldwide.

DETAILED DESCRIPTION:
This is a descriptive, mono-center study aimed at comparing a local triage score with that of qsofa in patients presenting to the Sahloul Emergency Department with sepsis.

A local triage score was calculated for each patient consulting the emergency room; this score makes it possible to classify patients according to severity and to predict the time to treatment.

A form is completed prospectively for each patient admitted to the observation unit whose diagnosis of sepsis is confirmed and validated by a senior during the morning staff.

The validated data were included in the ReSSUS register (Sepsis Register of the Sahloul Emergency Department). This is an observational database on the management of sepsis admitted to the emergency department in Sahloul. It ensures a high level of confidentiality and protection of medical data.

Subsequent follow-up of patients was done by telephone contact to verify mortality at one month and one year.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* each patient diagnosed as an acute Sepsi consulting the emergencies of CHU Sahloul, Sousse

Exclusion Criteria:

* no exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: each patient diagnosed as an acute Sepsi consulting the emergencies of CHU Sahloul, Sousse
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Mortality | one month

SECONDARY OUTCOMES:
Mortality and /or readmission | one year
  Mortality and /or readmission

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Boukef, professor, Principal Investigator — CHU Sahloul, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided